CLINICAL TRIAL: NCT03459820
Title: Differences in Optimal Prostate Cancer Patient Management as Proposed by a Panel of Experts Before and After 18F-DCFPyL PET/CT
Brief Title: Prostate Cancer Patient Management With 18F-DCFPyL PET/CT
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-002
Record Dates: First submitted 2018-03-03; First posted 2018-03-09 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL PET/CT (Experimental): 18F-DCFPyL PET/CT Scan
  Interventions: Diagnostic Test: 18F-DCFPyL PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-DCFPyL PET/CT — 18F-DCFPyL Positron Emission Tomography/Computed Tomography Scan

SUMMARY:
This is a multi-center, single-arm, open-label, phase III trial in patients with biopsy-proven prostate cancer. Patients will receive regular standard of clinical care. The only study-specific procedures will the administration of 18F-DCFPyL followed by a PET/CT scan. Differences in theoretical optimal clinical management based on a review of clinical, biochemical and radiographic subject data before and after 18F-DCFPyL PET/CT imaging by a central panel of experts will be captured at study completion.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to assess the differences in theoretical optimal clinical management afforded by 18F-DCFPyL PET/CT in prostate cancer patients as proposed by a central panel of experts.

Primary endpoint:

1. Differences in theoretical optimal clinical management based on a review of clinical, histopathological, biochemical and radiographic subject data both before and after 18F-DCFPyL PET/CT imaging retrospectively by a central panel of experts.

Secondary endpoints:

1. 18F-DCFPyL PET/CT scan positivity fraction in patients with biochemically recurrent prostate cancer, stratified by PSA.
2. Immediate AE up to 90 minutes post-administration of 18F-DCFPyL.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18 years or older
* Previously diagnosed with prostate cancer, under referring physician's care
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine (or prone) for up to 40 minutes and tolerating intravenous cannulation for injection

Cohort A - High risk staging (HRS): Staging of high risk not previously treated patients as defined by any one of the following:

* Gleason score > 7
* Serum PSA > 15 ng/ml
* T stage of T3 or greater on TNM staging
* Equivocal/inconclusive conventional staging such as CT, MRI or bone scan
* Clinical suspicion of advance stage disease (e.g. bone pain)

Cohort B - Biochemical recurrence: Restaging of biochemically recurrent prostate cancer patients as defined by increasing serum PSA on serial measurements and current PSA above 0.1 ng/ml following any treatment for prostate cancer.

Exclusion Criteria:

* Patients who are medically unstable (e.g. acute cardiac or respiratory distress or hypotensive)
* Patients who exceed the safe weight limit of the PET/CT bed (usually approximately 400 lbs.) or who cannot fit through the PET/CT bore (usually approximately 70 cm diameter)
* Patients with unmanageable claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with prostate cancer are included.
Enrollment: 1500 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Differences in optimal clinical management | 30 days
  Differences in theoretical optimal clinical management based on a review of clinical, histopathological, biochemical and radiographic subject data both before and after 18F-DCFPyL PET/CT imaging retrospectively by a central panel of experts.

SECONDARY OUTCOMES:
Scan positivity fraction in BCR by PSA. | 30 days
  18F-DCFPyL PET/CT scan positivity fraction in patients with biochemically recurrent prostate cancer, stratified by PSA.
Adverse events | 2 hours
  Immediate AE up to 90 minutes post-administration of 18F-DCFPyL.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided